CLINICAL TRIAL: NCT03016819
Title: A Phase III Study of AL3818 (Anlotinib, Catequentinib) Hydrochloride Monotherapy in Subjects With Metastatic or Advanced Alveolar Soft Part Sarcoma, Leiomyosarcoma and Synovial Sarcoma
Brief Title: Phase III Trial of Anlotinib, Catequentinib in Advanced Alveolar Soft Part Sarcoma, Leiomyosarcoma, Synovial Sarcoma (APROMISS)
Acronym: APROMISS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Advenchen Laboratories, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AL3818-US-004
Record Dates: First submitted 2017-01-06; First posted 2017-01-11 (Estimated); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Alveolar Soft Part Sarcoma; Leiomyosarcoma; Synovial Sarcoma; Soft-Tissue Sarcoma
MeSH Terms: conditions — Sarcoma, Alveolar Soft Part; Leiomyosarcoma; Sarcoma, Synovial; Sarcoma | interventions — anlotinib; Dacarbazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Indication D (Leiomyosarcoma, AL3818 vs placebo) of study AL3818-US-004 is double-blinded. Indications A (alveolar soft part sarcoma, single arm with AL3818), B (Leiomyosarcoma, AL3818 vs dacarbazine), C (Synovial sarcoma, AL3818 vs dacarbazine) are open-label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Indication A: ASPS AL3818 Arm - CLOSED (Experimental): All subjects with ASPS will be assigned to the open-label AL3818 arm to receive 12 mg AL3818 capsules orally once daily in 21-day cycles (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21).
  Interventions: Drug: AL3818
- Indication B: LMS AL3818 Arm - CLOSED (Experimental): Subjects with LMS will be randomized in a 2:1 ratio to receive either AL3818 or IV dacarbazine. Subjects randomized to AL3818 will receive 12 mg AL3818 capsules orally once daily in 21-day cycles (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21).
  Interventions: Drug: AL3818
- Indication B: LMS Dacarbazine Arm - CLOSED (Active Comparator): Subjects with LMS will be randomized in a 2:1 ratio to receive either AL3818 or IV dacarbazine. Subjects randomized to IV dacarbazine will receive dacarbazine at a dose of 1000 mg/m^2 as a 20-120 minute IV infusion on Day 1 of each 21-day treatment cycle.
  Interventions: Drug: Dacarbazine
- Indication C: SS AL3818 Arm - CLOSED (Experimental): Subjects with SS will be randomized in a 2:1 ratio to receive either AL3818 or IV dacarbazine. Subjects randomized to AL3818 will receive 12 mg AL3818 capsules orally once daily in 21-day cycles (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21).
  Interventions: Drug: Dacarbazine
- Indication C: SS Dacarbazine Arm - CLOSED (Active Comparator): Subjects with SS will be randomized in a 2:1 ratio to receive either AL3818 or IV dacarbazine. Subjects randomized to IV dacarbazine will receive dacarbazine at a dose of 1000 mg/m^2 as a 20-120 minute IV infusion on Day 1 of each 21-day treatment cycle.
  Interventions: Drug: Dacarbazine
- Indication D: LMS AL3818 or Placebo Arm - CLOSED (Placebo Comparator): Subjects with LMS will be randomized in a 2:1 ratio to receive either AL3818 or placebo in a double-blind manner. AL3818 or placebo will be administrated as one 12 mg capsule orally once daily in 21-day cycles for 14 days on treatment (Days 1-14) and 7 days off treatment (Days 15-21).
  Interventions: Drug: AL3818 or placebo

INTERVENTIONS:
Drug: AL3818 — Anlotinib (AL3818) 12 mg orally administered once daily in 21-day cycles (14 days on treatment, 7 days off treatment)
  Other Names: Catequentenib; Anlotinib
  Arms: Indication A: ASPS AL3818 Arm - CLOSED; Indication B: LMS AL3818 Arm - CLOSED
Drug: Dacarbazine — Dacarbazine 1000 mg/m2 as a 20-120 minute IV infusion on Day 1 of each 21-day treatment cycle
  Other Names: DTIC
  Arms: Indication B: LMS Dacarbazine Arm - CLOSED; Indication C: SS AL3818 Arm - CLOSED; Indication C: SS Dacarbazine Arm - CLOSED
Drug: AL3818 or placebo — AL3818 or placebo 12 mg orally administered once daily in 21-day cycles (14 days on treatment, 7 days off treatment)
  Arms: Indication D: LMS AL3818 or Placebo Arm - CLOSED

SUMMARY:
THIS STUDY IS CURRENTLY RECRUITING PATIENTS WITH ALVEOLAR SOFT PART SARCOMA ONLY AND IS NO LONGER RECRUITING PATIENTS WITH SYNOVIAL SARCOMA OR LEIOMYOSARCOMA.

This study evaluates the safety and efficacy of AL3818 (anlotinib) hydrochloride in the treatment of metastatic or advanced alveolar soft part sarcoma (ASPS), leiomyosarcoma (LMS), and synovial sarcoma (SS). All participants with ASPS will receive open-label AL3818. In participants with LMS or SS, AL3818 will be compared to IV dacarbazine. Two-thirds of the participants will receive AL3818, one-third of the participants will receive IV dacarbazine.

DETAILED DESCRIPTION:
THIS STUDY IS CURRENTLY RECRUITING PATIENTS WITH ALVEOLAR SOFT PART SARCOMA ONLY AND IS NO LONGER RECRUITING PATIENTS WITH SYNOVIAL SARCOMA OR LEIOMYOSARCOMA.

APROMISS is a phase 3 study evaluating the safety and efficacy of AL3818 (anlotinib) hydrochloride in the treatment of metastatic or advanced alveolar soft part sarcoma (ASPS), leiomyosarcoma (LMS), and synovial sarcoma (SS). Population pharmacokinetics and exploratory exposure-response analyses will also be conducted in subjects receiving AL3818.

Indication A: 56 subjects with metastatic or advanced ASPS not amenable to surgical resection will receive open-label AL3818 at a dose of 12 mg once daily in 21-day cycles (14 days on treatment, 7 days off treatment) until disease progression (defined by RECIST version 1.1) ot unacceptable toxicity. The primary endpoint is objective response rate (ORR), secondary endpoint is duration of response (DOR). - CLOSED

Indication B: 68 subjects with metastatic or advanced LMS who have failed at least one prior line of approved therapy will be enrolled and randomized in a 2:1 ratio to receive either AL3818 (12 mg once daily in 21-day cycles) or IV dacarbazine until disease progression (defined by RECIST version 1.1) or unacceptable toxicity. Subjects randomized to dacarbazine will have the option to crossover and receive AL3818 at the time of documented disease progression. The primary endpoint is progression free survival (PFS), the secondary endpoint is objective response rate (ORR). - CLOSED

Indication C: 95 subjects with with metastatic or advanced SS who have failed at least one prior line of approved therapy, including first-line anthracycline-containing chemotherapy, will be enrolled and randomized in a 2:1 ratio to receive either AL3818 (12 mg once daily in 21-day cycles) or IV dacarbazine until disease progression (defined by RECIST version 1.1) or unacceptable toxicity. Subjects randomized to dacarbazine will have the option to crossover and receive AL3818 at the time of documented disease progression. The primary endpoint is progression free survival (PFS), the secondary endpoint is objective response rate (ORR). - CLOSED

Indication D - LMS: 106 subjects with histologically proven, unresectable, recurrent, locally advanced or metastatic leiomyosarcoma (of soft tissue, cutaneous origin, and vascular origin who have failed at least one prior line of standard therapy (including anthracycline-based therapy) and are ineligible for or refuse standard second-line therapy or are suitable for third- and further-line treatment will be enrolled. Subjects will be randomized with a 2:1 ratio to receive either blinded AL3818 or placebo with approximately 71 subjects in the AL3818 group and 35 subjects in the placebo group until disease progression (defined by RECIST version 1.1) or unacceptable toxicity. Subjects randomized to placebo will have the option to crossover and receive AL3818 at the time of documented disease progression (and after crossover unblinding). The primary endpoint is progression free survival (PFS), the secondary endpoint is objective response rate (ORR). - CLOSED

ELIGIBILITY:
Inclusion Criteria

1. Written informed consent provided before any study-specific procedures are initiated. Subject must be able to understand and be willing to sign a written informed consent form.
2. Male or female at least 18 years of age.
3. a. Indication A - ASPS: Histologically proven, unresectable, locally advanced or metastatic alveolar soft part sarcoma. b. CLOSED Indication B - LMS: Histologically proven, unresectable, recurrent, locally advanced or metastatic leiomyosarcoma (of soft tissue, cutaneous origin, vascular origin and of the bone). c. CLOSED Indication C - SS: Histologically proven, unresectable, recurrent, locally advanced or metastatic synovial sarcoma. d. CLOSED Indication D - LMS: Histologically proven, unresectable, recurrent, locally advanced or metastatic leiomyosarcoma (of soft tissue, cutaneous origin, and vascular origin).
4. a. Indication A - ASPS: Subjects with or without prior therapy. b. Indications B - LMS: Subjects previously treated with at least one prior line of approved therapy. (New Recruitment Suspended) c. Indication C - SS: Subjects previously treated with at least one prior line of standard systemic therapy, including first-line anthracycline containing regimen (except if medically contraindicated or refused by subject). d. Indication D - LMS: Treatment of patients with metastatic or advanced leiomyosarcoma (LMS) who have failed at least one prior line of standard therapy and are ineligible for or refuse standard second-line therapy or are suitable for third- and further-line treatment. Patients must have received and progressed on prior therapy and have been treated any line with an anthracycline.
5. Show clinical or objective disease progression after the last administration of the last standard therapy or have stopped standard therapy due to intolerability within 6 months of enrollment (excluding ASPS subjects who have not received prior therapy).
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
7. Has measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 confirmed by CT or MRI scan of the chest, abdomen and pelvis (and other areas of disease) within 28 days prior to enrollment.
8. Life expectancy of at least 3 months.
9. Females of childbearing potential must have a negative pregnancy test (by serum beta- HCG) within 7 days prior to the start of treatment.
10. Female of childbearing potential must be surgically sterile (have had a hysterectomy or bilateral oophorectomy, tubal ligation), abstinent (at the discretion of the investigator), or agree to use adequate contraception since signing of the informed consent form until at least 3 months after the last study drug administration. Females of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 2 years. Males must agree to use adequate contraception since signing of the informed consent form until at least 3 months after the last study drug administration. Adequate contraception is defined in the study as any medically recommended method (or combination of methods) at the discretion of the investigator.
11. Adequate hematologic, hepatic and renal function as assessed by the following laboratory requirements conducted within 28 days of enrollment:

    1. Total bilirubin < the upper limit of normal (ULN), unless the patient has documented Gilbert's disease for which the total bilirubin should be < 3.
    2. Alanine aminotransferase and aspartate aminotransferase < 2.5 of the ULN (< 5 x of ULN for subjects with liver involvement of their cancer)
    3. Amylase and lipase < 1.5 x of ULN
    4. Serum creatinine < 1.5 x of ULN
    5. Glomerular filtration rate > 30ml/min/1.73 m2 according to the Modified Diet in Renal Disease abbreviated formula or creatinine clearance (CrCL) > 60 ml/min (Cockcroft and Gault) or by 24 hour urine collection.
    6. International normalize ratio (INR) and the activated partial thromboplastin time (aPTT/PTT) < 1.5 x ULN. (Subjects who are therapeutically treated with an agent such LMWH or heparin will be allowed to participate provided that no prior evidence of an underlying abnormality in coagulation parameters exists)
    7. Platelet count > 100,000 cells/mm3, hemoglobin > 9 g/dL, absolute neutrophil count > 1,500 cells/mm3
    8. Alkaline phosphatase limit <2.5 x ULN (<5 x ULN for subjects with liver involvement of their cancer)
    9. Urine protein < 30 mg/dL. If urine protein is > 30 mg/dL, a 24-hour urine collection will be required and must show total protein excretion <1,000 mg per 24 hours or spot urine protein (mg/dL) to creatinine (mg/dL) ratio must be <1.0.
12. Left ventricular ejection fraction (LVEF) of > 50% by ECHO or MUGA within 56 days of enrollment.
13. Two readings of systolic blood pressure < 140 mm Hg and diastolic blood pressure < 90 mm Hg at screening taken at least 5 minutes apart in the sitting position after 5 minutes of rest. Subjects with well managed hypertension who are on oral antihypertensives must be on their current medication(s) and stable dose(s) for at least 2 weeks prior to enrollment.

Exclusion Criteria

1. Prior treatment with or have known hypersensitivity to AL3818.
2. a. Indication A - ASPS: Prior treatment with cediranib. b. Indication B - LMS: Prior treatment with or have known hypersensitivity to dacarbazine. (New Recruitment Suspended) c. Indication C - SS: Prior treatment with or have known hypersensitivity to dacarbazine.

   d. Indication D - LMS: Prior treatment with anlotinib.
3. Previous or concurrent cancer that is distinct in primary site or histology from ASPS, LMS, or SS within 5 years before enrollment except for successfully treated in situ carcinoma, non-melanoma skin cancer and superficial bladder tumors (Ta, Tis and T1).
4. Received last dose of systemic cytotoxic therapy or investigational therapy within 21 days of enrollment or last dose of hormonal therapy, immunotherapy, targeted therapy or any other type of non-cytotoxic anti-cancer therapy within 14 days of enrollment.
5. Prior treatment with extended-field radiotherapy (EFRT) within 28 days of enrollment or prior treatment with any other form of radiotherapy within 14 days of enrollment.
6. Known active CNS metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided that they are stable with no evidence of progression by imaging, and all neurologic symptoms have returned to baseline, and should not be using corticosteroids for at least 7 days prior to study treatment.
7. Cavitary tumors or tumors invading or abutting large blood vessels in the thorax.
8. History of gastrointestinal perforation, abdominal fistula or intra-abdominal abscess within 6 months of enrollment.
9. Known history of bleeding disorders (e.g., von Willebrand disease or hemophilia).
10. Clinically significant bleeding such as gross hematuria, gastrointestinal bleeding and hemoptysis within 6 months prior to enrollment.
11. CTCAE version 4.03 > grade 2 pulmonary hemorrhage or > grade 3 of other forms of bleeding within 28 days prior to enrollment.
12. History of untreated deep venous thrombosis (DVT) within the past 6 months. Patients with recent DVT who are treated with therapeutic anti-coagulating agents (excluding therapeutic warfarin which is exclusionary) for at least 14 days prior to start of study treatment.
13. Use of aspirin (>325 mg/day) within 10 days prior to the first dose of study treatment.

    The use of prophylactic therapeutic anti-coagulants are allowed provided that INR or aPTT are within therapeutic limits (according to the medical standard of the enrollment institution) and patient has been on a stable dose of anticoagulants for at least two weeks prior to the first dose of study treatment.
14. Serious non-healing wound, active ulcer.
15. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to enrollment or minor surgical procedure within 7 days of enrollment.
16. CTCAE version 4.03 > grade 3 peripheral neuropathy
17. Any unrecovered toxicity reactions of CTCAE version 4.03 > grade 1 caused by any previous therapy (excluding alopecia and neurotoxicity < grade 2)
18. QTcF > 470 msec (per Fridericia's formula) on electrocardiogram within 28 days of enrollment.
19. Severe and uncontrolled disease, including:

    1. Class I and above myocardial ischemia or myocardial infarction, cardiac arrhythmia and Class 2 or above congestive heart failure classified according to New York Heart Association (NYHA)
    2. Active or failed to control serious infections (CTCAE version 4.03 > grade 2 infections)
    3. Liver disease such as cirrhosis of the liver, decompensated liver disease, chronic active hepatitis needing anti-viral therapy
    4. Renal failure needing hemodialysis or peritoneal dialysis
    5. Poorly controlled diabetes (HgA1C >8)
    6. Untreated and uncontrolled epileptic seizures
    7. History of psychotropic drug abuse and inability to quit
    8. Untreated psychiatric disorders
20. Known HIV-positive
21. Had organ transplantation
22. Clinical conditions affecting the intake and use of oral medications (e.g., inability to swallow, chronic diarrhea, and intestinal obstruction)
23. Females who are pregnant or are breast-feeding.
24. Concomitant treatment with strong inhibitors or inducers of CYP1A2, CYP3A4 or CYP3A5; or sensitive substrates with narrow therapeutic index (TI) of CYP3A4, CYP2C9 and CYP2C19; or QT prolongating medications within 14 days prior to enrollment and during the study unless there was an emergent or life-threatening medical condition that required it.
25. Any medical intervention, condition or any other circumstance which in the opinion of the investigator or the sponsor's medical monitor, could compromise adherence to study procedures or study objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Estimated)
Dates: Start 2017-08-15 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) (ASPS) | Up to 48 months
  To determine ORR in subjects with ASPS, defined as percentage of subjects who achieve a Complete Response (CR) or Partial Response (PR) as best responses according to RECIST 1.1 as evaluated by a blinded independent radiological review (BICR).
Progression Free Survival (PFS) (LMS/SS) | From time of randomization to the date of disease progression or death from any cause, up to 48 months
  To compare PFS in subjects with LMS or SS randomized to AL3818 versus dacarbazine, defined a median number of months from the date of randomization until the first documented sign of disease progression or death due to any causes, whichever occurs earlier as evaluated by a blinded independent radiologic review (BICR).

SECONDARY OUTCOMES:
Duration of Response (DOR) (ASPS) | Up to 48 months
  To determine DOR in subjects with ASPS, defined as median number of months from date of first documented objective response until first documented sign of disease progression or death due to any causes
Objective Response Rate (ORR) (LMS/SS) | Up to 48 months
  To compare ORR in subjects with LMS or SS randomized to AL3818 versus dacarbazine, defined as percentage of subjects who achieve a Complete Response (CR) or Partial Response (PR) as best responses according to RECIST 1.1 as evaluated by a blinded independent radiological review (BICR).

CONTACTS AND LOCATIONS:
Overall Officials: Paul CEO, Study Director — Advenchen Laboratories, LLC
Locations (23):
- United States (16):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - University of California Los Angeles, Los Angeles, California
  - Sarcoma Oncology Center, Santa Monica, California
  - Stanford Medicine Cancer Institute, Stanford, California
  - University of Colorado Denver, Aurora, Colorado
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Northwestern University, Chicago, Illinois
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University St. Louis, St Louis, Missouri
  - Thomas Jefferson Hospital - Sidney Kimmel Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - UW Medicine-Seattle Cancer Care Alliance, Seattle, Washington
- China (2):
  - Beijing Cancer Hospital, Beijing
  - Shanghai Sixth People's Hospital, Shanghai
- Italy (3):
  - Istituto Nazionale dei Tumori, Milan
  - University of Palermo, Palermo
  - University Campus Bio-Medico, Rome
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain
- Royal Marsden Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No